CLINICAL TRIAL: NCT00002882
Title: Adjuvant Therapy for Melanoma Patients With Regional Lymph Node Metastases With Interferon Alfa-2B vs. Biochemotherapy Using Cisplatin + Vinblastine + DTIC + Interferon Plus IL-2
Brief Title: Interferon Alfa With or Without Combination Chemotherapy Plus Interleukin-2 in Treating Patients With Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID95-196; P30CA016672 (NIH); MDA-ID-95196 (Other: UT MD Anderson Cancer Center); MDA-DM-95196 (Other: UT MD Anderson Cancer Center); NCI-G96-1089; CDR0000065188 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Melanoma; Skin Cancer
Keywords: stage III melanoma
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — aldesleukin; Interleukin-2; Interferon-alpha; Interferon alpha-2; Cisplatin; Dacarbazine; Vinblastine; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IFN-A Therapy Schedule A (Experimental): Schedule A: IV Interferon alfa-2b (IFN-A) induction 5 times a week for 4 weeks followed by subcutaneous IFN-A maintenance 3 times a week for 48 weeks.
  Interventions: Biological: Recombinant Interferon Alfa (IFN-A)
- IFN-A Therapy Schedule B (Experimental): Schedule B: Subcutaneous IFN-A 3 times a week for 52 weeks.
  Interventions: Biological: Recombinant Interferon Alfa (IFN-A)
- Adjuvant Biochemotherapy (Experimental): Cisplatin IV Days 1-4; Vinblastine IVPB Days 1-4; Dacarbazine (DTIC) IVPB on Day 1; IFN-A is given subcutaneously on days 1-5; IL-2 continuous infusion for 96 hours on Days 1-4. Each course repeated every 21 days for 4 courses.
  Interventions: Biological: Aldesleukin (IL-2); Biological: Recombinant Interferon Alfa (IFN-A); Drug: Cisplatin; Drug: Dacarbazine; Drug: Vinblastine; Procedure: Adjuvant Therapy

INTERVENTIONS:
Biological: Aldesleukin (IL-2) — Infusion for a total of 96 hours on days 1-4
  Other Names: IL-2; Interleukin-2; Proleukin
  Arms: Adjuvant Biochemotherapy
Biological: Recombinant Interferon Alfa (IFN-A) — IFN-A Therapy Groups:
  Schedule A: IV IFN-A induction 5 times a week for 4 weeks followed by subcutaneous IFN-A maintenance 3 times a week for 48 weeks.
  Schedule B: Subcutaneous IFN-A 3 times a week for 52 weeks
  Adjuvant Biochemotherapy Group: IFN-A is given subcutaneously on days 1-5
  Other Names: interferon alfa-2b; IFN-A
Drug: Cisplatin — IV Days 1-4
  Other Names: CDDP; Platinol; Platinol-AQ
  Arms: Adjuvant Biochemotherapy
Drug: Dacarbazine — IVPB on day 1
  Other Names: DTIC
  Arms: Adjuvant Biochemotherapy
Drug: Vinblastine — IVPB on days 1-4
  Other Names: Velban
  Arms: Adjuvant Biochemotherapy
Procedure: Adjuvant Therapy — Patients receiving adjuvant radiotherapy will start adjuvant systemic therapy within 8 weeks from lymphadenectomy and a week after completion of and recovery from radiotherapy.
  Arms: Adjuvant Biochemotherapy

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells. Interleukin-2 may stimulate a person's white blood cells to kill melanoma cells. It is not yet known whether interferon alfa plus combination chemotherapy and interleukin-2 is more effective than interferon alfa alone in treating patients with melanoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of interferon alfa with or without combination chemotherapy plus interleukin-2 in treating patients with melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of postoperative adjuvant therapy with interferon alfa-2b (IFN-A) administered subcutaneously with or without IV induction vs concurrent biochemotherapy including cisplatin, vinblastine, DTIC, IFN-A and IL-2 and in melanoma patients with regional lymph node metastases that have been surgically resected.
* Determine the relative toxic effects associated with adjuvant therapy with IFN-A and concurrent biochemotherapy including cisplatin, vinblastine, DTIC, IFN-A, and IL-2 and their effect on the quality of life.
* Determine the prognostic value of detection of melanoma cells in the peripheral blood using RT/PCR for tyrosinase mRNA.

OUTLINE: This is a randomized study. All patients are stratified according to prognostic factors.

Patients are randomly allocated to 1 of 2 treatment options. Treatment 1 uses interferon alfa-2b (IFN-A) therapy, and treatment 2 includes adjuvant biochemotherapy.

Patients who are randomized to IFN-A will be further stratified and randomized to one of two interferon schedules.

* Schedule A: IV IFN-A induction 5 times a week for 4 weeks followed by subcutaneous IFN-A maintenance 3 times a week for 48 weeks.
* Schedule B: Subcutaneous IFN-A 3 times a week for 52 weeks. Adjuvant biochemotherapy begins immediately after registration on the study. Cisplatin is given IV on days 1-4; vinblastine is given IVPB on days 1-4; dacarbazine (DTIC) is given IVPB on day 1; IFN-A is given subcutaneously on days 1-5; IL-2 is given by continuous infusion for a total of 96 hours on days 1-4. Each course of therapy is repeated every 21 days for 4 courses. Patients receiving adjuvant radiotherapy will start adjuvant systemic therapy within 8 weeks from lymphadenectomy and a week after completion of and recovery from radiotherapy.

PROJECTED ACCRUAL: A total of 200 patients (100 patients in each arm) will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically diagnosed malignant melanoma with regional lymph node metastases
* Undergone complete lymph node dissection and free of any residual tumor
* No greater than 90 days from diagnosis of regional lymph nodes metastases
* No distant or resected in-transit metastases

PATIENT CHARACTERISTICS:

Age:

* 10 to 66
* 66 to 70 if in excellent physical condition

Performance status:

* 0-2

Life expectancy:

* At least 12 months

Hematopoietic:

* Hemoglobin greater than 10 g/dL
* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.2 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Other:

* No serious intercurrent illness that would compromise tolerance of therapy and long term survival
* Must be able to participate in follow up for minimum of 5 years
* No second malignancy except:

  * In situ cervical cancer
  * Basal or squamous skin cancer
* Must be able to physically and emotionally tolerate biochemotherapy
* No history of pulmonary or cardiac dysfunction, e.g., cardiac rhythm disturbance, congestive heart failure, coronary bypass, or impaired cardiac ejection fraction

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy with interferon or IL-2
* No concurrent immunomodulators

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No concurrent steroids

Radiotherapy:

* Prior adjuvant local radiotherapy allowed for head and neck

Surgery:

* No greater than 8 weeks after definitive surgery for lymph node metastases

Other:

* No concurrent nonsteroid anti-inflammatory drugs, or other prostaglandin synthetase inhibitors

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 1995-11; Primary Completion 2003-08 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Interferon Alfa with/without Combination Chemotherapy + Interleukin-2 for Melanoma | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Agop Y. Bedikian, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Kim KB, Legha SS, Gonzalez R, Anderson CM, Johnson MM, Liu P, Papadopoulos NE, Eton O, Plager C, Buzaid AC, Prieto VG, Hwu WJ, Frost AM, Alvarado G, Hwu P, Ross MI, Gershenwald JE, Lee JE, Mansfield PF, Benjamin RS, Bedikian AY. A randomized phase III trial of biochemotherapy versus interferon-alpha-2b for adjuvant therapy in patients at high risk for melanoma recurrence. Melanoma Res. 2009 Feb;19(1):42-9. doi: 10.1097/CMR.0b013e328314b84a. PMID 19430405
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org